CLINICAL TRIAL: NCT06352450
Title: Comparison of Active Isolated Stretching Versus Myofascial Release of Knee Joint in Office Workers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DPT/Batch-Fall19/558
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Stiffness; Spine; Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active isolated stretching (AIS) (Experimental)
  Interventions: Diagnostic Test: Active isolated stretching (AIS)
- Myofascial release (MFR) (Experimental)
  Interventions: Diagnostic Test: Myofascial release (MFR)

INTERVENTIONS:
Diagnostic Test: Active isolated stretching (AIS) — Active isolated stretching (AIS) is a technique that involves stretching specific muscles or muscle groups while actively engaging the opposing muscles. It typically involves holding a stretch for 1-2 seconds and then releasing. This method aims to improve flexibility, increase range of motion, and enhance muscle function.
  Other Names: AIS
  Arms: Active isolated stretching (AIS)
Diagnostic Test: Myofascial release (MFR) — Myofascial release (MFR) is a technique used to release tension and tightness in the fascia, which is the connective tissue that surrounds and supports muscles and organs. It involves applying gentle, sustained pressure to specific areas of the body to help relax the fascia and alleviate restrictions. MFR aims to improve mobility, reduce pain, and enhance overall movement and function.
  Other Names: MFR
  Arms: Myofascial release (MFR)

SUMMARY:
"Office workers often spend long hours sitting, which can lead to stiffness and reduced mobility. By studying these two techniques AIS and MFR, we can determine which one is more effective in helping office workers to improve their flexibility and range of motion in the knee joint because their sedentary work environment often leads to musculoskeletal issues, including limited knee joint mobility.

AIS involves stretching specific muscles while actively engaging opposing muscles to enhance the effectiveness of the stretch. It aims to increase the extensibility of muscles and improve joint mobility. On the other hand, MFR focuses on releasing tension and adhesions in the fascia, the connective tissue surrounding muscles and joints, to restore mobility and reduce pain.

Understanding the benefits and effectiveness of these techniques will contribute to evidence-based practices in occupational health and help office workers maintain optimal joint health"

DETAILED DESCRIPTION:
"Office workers often spend long hours sitting, which can lead to stiffness and reduced mobility. By studying these two techniques AIS and MFR, we can determine which one is more effective in helping office workers to improve their flexibility and range of motion in the knee joint because their sedentary work environment often leads to musculoskeletal issues, including limited knee joint mobility.

AIS involves stretching specific muscles while actively engaging opposing muscles to enhance the effectiveness of the stretch. It aims to increase the extensibility of muscles and improve joint mobility. On the other hand, MFR focuses on releasing tension and adhesions in the fascia, the connective tissue surrounding muscles and joints, to restore mobility and reduce pain.

Understanding the benefits and effectiveness of these techniques will contribute to evidence-based practices in occupational health and help office workers maintain optimal joint health"

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects with age group between 25 to 45 years with prolonged sitting 2. both males and females will be included. 3. Patients with diagnosed with reduced hamstrings flexibility and range of motion which we checked by doing walking (normal ranges 0 to 60 in flexion and 0 to 10 in extension) and squatting (normal range when knees bend to angle of 90 to 120 in flexion and 0 in extension) 4. Patients with reduced straight leg raise. 5. Patients with pain in posterior compartment of thigh 6. Asymptomatic patients will be included. 7. Patients with restricted mobility of lower limb due to Hamstring shortness. 8. Symptomatic patients with hamstring tightness like of low back pain, pelvic tightness, knee osteoarthritis (grade 1 and 2) are included in the research.

Exclusion Criteria:

* 1. Patients with prolapsed disc will excluded. 2. Patients with lower extremity injuries (strain, sprain, ligament injuries, etc.) in last 6 months will be excluded.

  3. Patients with severe hamstring injury either acute or chronic will be excluded.

  4. Patients with visual acute swelling in the region of hamstring muscle 5. Patients with fracture of any type and area. 6. Patients with dislocations or subluxations present will be excluded. 7. Patient recommended for TKR of knee joint. 8. Patients with any neurological disease like lumbar/cervical herniation, polyneuropathy, scoliosis etc.) 9. Patient with any tumor of hip or knee with traumatic brain injury, spinal cord injuries will be excluded

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Numaric Pain Scale | 6 Month
  Pain in office workers(Numaric Pain Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahra Medical complex Johar town, Laser spine center Model town, Laser spine center Johar town., Lahore, Pakistan